CLINICAL TRIAL: NCT01566669
Title: A Multicenter, Randomised, Double-blinded, Placebo-controlled Trial Comparing the Efficacy and Safety of Intravenous Parecoxib Sodium on Morphine Patient-controlled Epidural Analgesia After Gynecologic Surgery
Brief Title: Efficacy and Safety of Parecoxib on Morphine Patient-controlled Epidural Analgesia (PCEA) After Gynecologic Surgery
Acronym: PCEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Weifeng (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor-Investigator, Liu Weifeng, attending doctor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCEA
Record Dates: First submitted 2012-03-18; First posted 2012-03-29 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Benign Female Reproductive System Neoplasm
Keywords: Cyclooxygenase inhibitors; Morphine; Analgesia; patient-controlled; Gynecologic surgical procedures
MeSH Terms: conditions — Agnosia | interventions — parecoxib; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Before incision, patients in controlled Group received NS
  Interventions: Drug: Normal saline
- parecoxib sodium (Experimental): Before incision, parecoxib patients received 40mg of parecoxib IV
  Interventions: Drug: Parecoxib Sodium

INTERVENTIONS:
Drug: Parecoxib Sodium — Before incision, patients in Group P (n = 120) receive 40mg of parecoxib IV. Thereafter, parecoxib patients receive 40mg of parecoxib IV every 12 h for 48 h. 30 min before the end of surgery, a mixture of 6 mL of ropivacaine 0.25% and 2mg morphine was given epidurally. Epidural patient-controlled analgesia was initiated by using ropivacaine 0.125% (1.25 mg/ml) and morphine 0.005% (0.05 mg/ml) with a basal infusion rate of 2 ml/h, a demand dose of 2 ml, and a 15-min lockout.
  Other Names: Dynastat
  Arms: parecoxib sodium
Drug: Normal saline — Before incision, patients in Group C (n = 120) receive 2 mL of normal saline IV. Thereafter, they receive 2 mL of normal saline IV every 12 h for 48 h. 30 min before the end of surgery, a mixture of 6 mL of ropivacaine 0.25% and 2mg morphine was given epidurally. Epidural patient-controlled analgesia was initiated by using ropivacaine 0.125% (1.25 mg/ml) and morphine 0.005% (0.05 mg/ml) with a basal infusion rate of 2 ml/h, a demand dose of 2 ml, and a 15-min lockout.
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to determine the effects of parecoxib in combination with epidural morphine in providing analgesia for patients undergoing gynecological surgery.

DETAILED DESCRIPTION:
Researches have showed that the use of epidural and spinal block resulted in significant reduction in morbidity and mortality after surgery. Moreover, appropriate pain management results in better outcomes. Opioids therapy is recommended as the first choice medication for the management of postoperative pain but is associated with a number of undesirable adverse effects. A multimodal therapy for providing postoperative analgesia has advantages over the use of opioids alone. The use of NSAIDs and opioids together often improves analgesia and reduces the need for opioids in the postoperative period. Often, the combination of COX-2 inhibitors with epidural analgesia is preferred. With epidural analgesia, addition of COX-2 inhibitors may improve the analgesia and decrease the undesirable side effects.

ELIGIBILITY:
Inclusion Criteria:

* women scheduled for elective gynecological surgery under combined spinal-epidural anesthesia

Exclusion Criteria:

* contraindications for CSE placement
* known allergy, sensitivity, or contraindication to opioid and nonopioid analgesic drugs
* history of bleeding disorders, peptic ulceration, or anticoagulant use within the past month
* current pregnancy or breastfeeding
* history of known or suspected drug abuse
* unable to understand the use of pain assessment scales and the PCA device
* Patient with asthma or bronchospasm, requiring treatment with glucocorticoids
* poorly controlled hypertension or diabetes, a chronic or acute renal or hepatic disorder, or inflammatory bowel disease
* patients had taken antidepressants, narcotic analgesics, antihistamines, anxiolytics, hypnotics, sedatives, NSAIDs, or corticosteroids up to 24 h before receipt of the study medication

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
morphine-sparing effect of parecoxib | within 48 h after skin closure
  The primary end-point of this study was to quantify the morphine-sparing effect of a multimodal approach containing parecoxib compared with the standard PCEA approach in patients undergoing abdominal hysterectomy.

SECONDARY OUTCOMES:
pain intensity and side effects accompanied with PCEA and parecoxib | within 48 h after skin closure
  The secondary outcome included pain intensity, the patients' global evaluation, and side effects accompanied with PCEA and parecoxib, such as nausea, vomiting, pruritus, sedation, motor block in the lower extremities, and the time to passage of flatus and first bowel movement.Blood loss, length of hospitalization, and postoperative cardiovascular (CV) events were also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wenqi Huang, postgraduate, Study Chair — The First Affliated Hospital, Sun Yet-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu WF, Shu HH, Zhao GD, Peng SL, Xiao JF, Zhang GR, Liu KX, Huang WQ. Effect of Parecoxib as an Adjunct to Patient-Controlled Epidural Analgesia after Abdominal Hysterectomy: A Multicenter, Randomized, Placebo-Controlled Trial. PLoS One. 2016 Sep 13;11(9):e0162589. doi: 10.1371/journal.pone.0162589. eCollection 2016. PMID 27622453